CLINICAL TRIAL: NCT02702830
Title: Understanding Exercise Intolerance After Treatment for Cancer
Brief Title: MRI and Cardio-Pulmonary Exercise Testing in Evaluating Exercise Intolerance in Patients With Stage I-III Breast Cancer After Chemotherapy Treatment
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00036572; NCI-2016-00205 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 01915A (Other: Comprehensive Cancer Center of Wake Forest University); P30CA012197 (NIH)
Record Dates: First submitted 2016-03-01; First posted 2016-03-09 (Estimated); Last update posted 2019-04-26 (Actual); Status verified 2018-07

CONDITIONS: Healthy Subject; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage IIA Breast Cancer; Stage IIB Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Exercise Test; Clostridium perfringens epsilon-toxin; Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Diagnostic (MRI and CPET): Patients undergo CPET using a one-way breathing mask in 2 separate days 1-2 weeks apart. Patients also undergo MRI before and within 60 seconds after exercising.
  Interventions: Other: Cardiopulmonary Exercise Testing; Device: Magnetic Resonance Imaging

INTERVENTIONS:
Other: Cardiopulmonary Exercise Testing — Undergo CPET
  Other Names: CPET; CPX
Device: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging

SUMMARY:
This pilot research trial studies magnetic resonance imaging (MRI) and cardio (heart)-pulmonary (lung) exercise testing in evaluating exercise intolerance in patients with stage I-III breast cancer after treatment with chemotherapy drugs called anthracyclines. Anthracyclines are related with heart problems, cardiac abnormalities, bone and muscle dysfunction. Patients with breast cancer who are exposed to anthracycline drugs may also experience progressive fatigue and exercise intolerance which may limit daily activities and is an important barrier for patients returning to work. Using MRI and cardio-pulmonary exercise testing (CPET) may help doctors understand the causes of fatigue and exercise intolerance in patients receiving anthracycline chemotherapy and this may also allow doctors to plan better treatments to protect patients' heart, cardiovascular system, bone and muscle function.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility of performing upright treadmill cardio-pulmonary exercise stress testing utilizing magnetic resonance imaging.

II. To determine the reproducibility of measures of peak oxygen uptake (V02) and cardiac output as well as arterio-venous oxygen difference (A-V02) difference in survivors of breast cancer treatment and control participants.

OUTLINE:

Patients undergo CPET using a one-way breathing mask in 2 separate days 1-2 weeks apart. Patients also undergo MRI before and within 60 seconds after exercising.

ELIGIBILITY:
Inclusion Criteria:

* Women with stage I-III breast cancer who began their cancer treatment 1-2 years prior to this study and have received anthracycline based chemotherapy
* Women matched to age with our 16 post-cancer treatment participants

Exclusion Criteria:

* Those with contraindications for MRI such as ferromagnetic cerebral aneurysm clips or other intracranial metal, pacemakers, defibrillators, functioning neurostimulator devices or other implanted electronic devices
* Those with contraindications for exercise tolerance test (ETT) testing, including unstable angina or inability to exercise on a treadmill or stationary cycle
* Those who are pregnant, claustrophobic, or unable to provide informed consent

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult women with breast cancer or age-matched control
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2016-08-25 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
A-VO2 differences | Baseline to up to 2 weeks
  Descriptive statistics will be estimated for each measure at each of the two times they are measured. Correlation between the two assessments of each measure will be estimated and then establish a 95% confidence interval for this correlation. Difference between each assessment will be calculated and a 95% confidence interval for this difference will be estimated. A paired t-test will be performed to determine if the groups have a mean difference close to zero. The ratio of the variances for each measure at each time point will be examined. The ratio will be examined whether it is close to 1.0

CONTACTS AND LOCATIONS:
Overall Officials: William Hundley, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States